CLINICAL TRIAL: NCT06680713
Title: Effects of a Single Maximal Exercise Session on the Metabolic Function of Physically Inactive Young Adults
Brief Title: Single Maximal Exercise Session and the Metabolic Response of Physically Inactive Young Adults (EASY-Study)
Acronym: EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sergio Martinez-Huenchullan (Other)
Collaborators: Universidad Austral de Chile (Other)
Responsible Party: Sponsor-Investigator, Sergio Martinez-Huenchullan, Associate Professor, Universidad San Sebastián
Organization: Universidad San Sebastián (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-01; SOCHED 2023-01 (Other: Sociedad Chilena de Endocrinología y Diabetes)
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Physical Deconditioning
Keywords: Insulin; Metabolism; Exercise
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Progressive exercise test (Experimental): The incremental effort test will be performed. Thus, on a cycle ergometer, each participant will begin the test with a pedaling cadence of 60-70 RPM at 30W load. Every 3 minutes, this load will increase by 30W, always maintaining the same pedaling cadence. Heart rate, blood pressure, rating of perceived effort, pulse oximetry and muscle oximetry will be monitored throughout the test.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Progressive exercise testing on a cyclo ergometer

SUMMARY:
The goal of this clinical trial is to learn how the metabolic parameters of physically inactive young adults respond to a progressive exercise testing. The main questions it aims to answer are:

Does a progressive exercise test induce metabolic adaptations that differ from a normal or physiologic status? Does the changes in circulating insulin might indicate metabolic dysfunctions in physically inactive young adults? Researchers will compare the metabolic status at baseline (rest) and the responses immediately after the finalization of a progressive exercise test until fatigue by collecting blood and urine samples before and after the exercise testing.

Participants will:

Undergo a progressive exercise test on a cycle ergometer where vital signs such as heart rate, blood pressure, rating of perceived effort, pulse and muscle oximetry will be recorded during the test.

Visit the laboratory once where all procedure will be conducted there. Stay in touch for the following week in case some exercise-related symptoms develops.

DETAILED DESCRIPTION:
Design: This is a quasi-experimental study comparing pre-and post-intervention. The research question investigates the influence of changes in blood lactate influenced by exercise on the plasma concentration of FGF21 in physically inactive people. This project has the approval of the Scientific Ethics Committee of the Valdivia Health Service (Ord. 222/2022) and has Biosafety certification by the Institutional Biosafety Committee of the Austral University of Chile (No. 36/23).

Sample: People over 18 years of age (and up to 30 years of age) enrolled in the Physical Therapy program at the Austral University of Chile will be included. They must be physically inactive (perform less than 150 minutes/week of moderate physical activity and/or 75 minutes/week of vigorous physical activity) and without medical contraindications to perform physical activity. People who are taking medications that influence blood glucose or insulin levels and/or with anti-inflammatory effects will be excluded. The sample size calculation was performed considering the following parameters: a power of 95%, an alpha value of 0.05, a difference in pre- and post-intervention means of FGF21 of 50 pg/ml (100 vs 150 pg/ml), with a standard deviation for both groups of 50 pg/ml. With these data, the sample size is 16 participants, and considering a 20% drop-off, the final size is 20 participants, where recruitment will be by convenience and maintaining gender parity.

Variables: At the time of entering the study, the age years, and sex of the participants will be recorded. Anthropometric variables such as weight in kilograms and height in meters will be recorded using a scale (InBody® 270) and a height rod (SECA) respectively. From these measurements, the body mass index (BMI) will be calculated in kilograms/meters. For the calculations of the waist-hip ratio (WHR) and waist-height ratio (WHR), the waist circumference will be measured in centimeters using the navel area as a reference point. The hip circumference will be measured as the largest circumference obtained at the trochanteric femoral level. The levels of total and segmental muscle and fat mass will be measured using the InBody® 270 bioimpedance meter. The level of spontaneous physical activity will be measured using the International Physical Activity Questionnaire (IPAQ) in its short version. To induce elevations in blood lactate, an incremental load test will be applied on a cycle ergometer or stationary bicycle, in which the pedaling load will be increased by 30W every 3 minutes, starting from an initial load of 30W until reaching the point of fatigue. Before starting the test, participants will remain seated for 10 minutes, during which time heart rate, subjective sense of exertion (SSE) with the modified Borg Scale, blood pressure, pulse oximetry, and muscle (vastus lateralis of quadriceps) will be recorded at rest. In addition, a venous blood sample will be taken in a 2 ml tube with EDTA and another tube without anticoagulant for the subsequent plasma measurement of FGF21 with a specific ELISA kit for this (RayBio® catalog ELH-FGF21) and complementary biochemical tests (glycemia, insulinemia, total cholesterol, triglycerides, HDL, LDL, VLDL, non-HDL cholesterol, transaminases (GOT and GPT), creatinine, uric acid, urea and urea nitrogen). In addition, lactate measurement will be performed from a digital prick with a sterile lancet. For this, a specific reactive strip will be used, which will be measured with the AccuTrend Plus ® device. In parallel, the participant will be asked to bring a urine sample from the same day on an empty stomach for biochemical analysis (proteinuria, creatinuria, albuminuria, glucosuria). Once these measurements have been taken at rest, the incremental stress test will begin. Thus, on a cycle ergometer, each participant will begin the test with a pedaling cadence of 60-70 RPM at 30W load. Every 3 minutes this load will increase by 30W, always maintaining the same pedaling cadence. During the execution of the test, participants will always be supervised and guided by a professional physical therapist. Heart rate, pulse and muscle oximetry, and SSE will be assessed minute by minute, while blood pressure will be measured every 3 minutes. At the end of the test, the test execution time, the distance traveled in meters, heart rate, blood pressure, SSE, and final pulse and muscle oximetry will be recorded. The percentage of frequency reserve used during the test will be calculated with the Karvonen formula, which depends on the heart rates at rest and post-test. Fatigue at the end of the test will be understood as the fulfillment of one or more of the following criteria: use of heart rate reserve ≥ 90%, subjective feeling of effort ≥ 18/20 according to the original Borg scale, blood pressure ≥ 200/100 mg of Hg, the desire of the participant to finish the test (Figure 3).

Immediately after the test, a new venous blood sample will be taken in a 2 ml EDTA tube and another tube without anticoagulant. In addition, the post-exercise blood lactate concentration will be measured by finger prick using a specific reagent strip and with the AccuTrend Plus ® device. In addition, a post-exercise urine sample will be requested for the biochemical analysis previously described. Subsequently, the participant's vital signs will be monitored for 10 minutes after the test to ensure proper recovery.

It is reiterated that, as an assessment of potential confounding/intermediate variables, the following biochemical parameters will be measured from blood samples taken pre- and post-exercise: Total cholesterol, triglycerides, HDL, LDL, VLDL, non-HDL cholesterol, insulin, glucose, and transaminases (GOT, GPT), creatinine, uric acid, urea, and urea nitrogen. While, for urine samples, the levels of proteinuria, albuminuria, creatinuria, and glucose will be assessed.

Statistical analysis

Quantitative variables will be expressed as median and interquartile range, while qualitative variables will be described in terms of absolute frequencies. To calculate potential differences between pre-and post-stress test values, particularly lactate and FGF21, as well as transaminase levels and kidney function markers, the Wilcoxon test or Student t-test for related samples will be used, depending on how the data distribution behaves (normal or nonparametric). In addition, associations between lactate and FGF21 concentrations, both pre-and post-exercise, will be explored using the Spearman correlation index and bivariate regression models. In addition, other potential associations of interest will be explored using the Spearman correlation index. For all analyses, a p-value equal to or less than 0.05 will be considered statistically significant, using SPSS version 20 and GraphPad version 8 software.

ELIGIBILITY:
Inclusion Criteria:

* Physically inactive (less than 150 minutes of weekly moderate-intensity or less than 75 minutes of weekly vigorous physical activity.

Without medical contraindication to perform physical activity

Exclusion Criteria:

* Consumption of drugs with anti-inflammatory and/or hypoglycemic effects during the last two weeks.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Glycemia | Up to 2 months
  Glucose in mg/dl
Insulinemia | Up to 2 months
  Insulin in uUI/ml

SECONDARY OUTCOMES:
Total cholesterol | Up to 2 months
  Total cholesterol in mg/dl
HDL cholesterol | Up to 2 months
  HDL cholesterol in mg/dl
LDL cholesterol | Up to 2 months
  LDL cholesterol in mg/dl
VLDL cholesterol | Up to 2 months
  VLDL cholesterol in mg/dl
Triglycerides | Up to 2 months
  Triglycerides in mg/dl
GOT (transaminase) | Up to 2 months
  GOT in U/L
GPT (transaminase) | Up to 2 months
  GPT in U/L
Proteinuria | Up to 2 months
  Proteinuria in mg/dl
Creatinine clearance | Up to 2 months
  Creatinine clearance in g/L
Albuminuria | Up to 2 months
  Albuminuria in mg/L
Glucosuria | Up to 2 months
  Glucosuria in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Sergio F Martinez-Huenchullan, PhD, Principal Investigator — Universidad San Sebastián
Locations (1):
- Universidad San Sebastián, Valdivia, Los Ríos Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 30-10-2024 to 30-10-2026
Access Criteria: Data will be shared by contacting the principal investigator at sergio.martinez@uss.cl

REFERENCES:
- [Background] Goodwin ML, Harris JE, Hernandez A, Gladden LB. Blood lactate measurements and analysis during exercise: a guide for clinicians. J Diabetes Sci Technol. 2007 Jul;1(4):558-69. doi: 10.1177/193229680700100414. PMID 19885119
- [Background] Garneau L, Parsons SA, Smith SR, Mulvihill EE, Sparks LM, Aguer C. Plasma Myokine Concentrations After Acute Exercise in Non-obese and Obese Sedentary Women. Front Physiol. 2020 Feb 18;11:18. doi: 10.3389/fphys.2020.00018. eCollection 2020. PMID 32132925
- [Background] Slusher AL, Whitehurst M, Zoeller RF, Mock JT, Maharaj M, Huang CJ. Attenuated fibroblast growth factor 21 response to acute aerobic exercise in obese individuals. Nutr Metab Cardiovasc Dis. 2015 Sep;25(9):839-845. doi: 10.1016/j.numecd.2015.06.002. Epub 2015 Jun 16. PMID 26141939
- [Background] Sabaratnam R, Pedersen AJT, Kristensen JM, Handberg A, Wojtaszewski JFP, Hojlund K. Intact regulation of muscle expression and circulating levels of myokines in response to exercise in patients with type 2 diabetes. Physiol Rep. 2018 Jun;6(12):e13723. doi: 10.14814/phy2.13723. PMID 29924476
- [Background] Ming AY, Yoo E, Vorontsov EN, Altamentova SM, Kilkenny DM, Rocheleau JV. Dynamics and Distribution of Klothobeta (KLB) and fibroblast growth factor receptor-1 (FGFR1) in living cells reveal the fibroblast growth factor-21 (FGF21)-induced receptor complex. J Biol Chem. 2012 Jun 8;287(24):19997-20006. doi: 10.1074/jbc.M111.325670. Epub 2012 Apr 20. PMID 22523080
- [Background] Fisher FM, Maratos-Flier E. Understanding the Physiology of FGF21. Annu Rev Physiol. 2016;78:223-41. doi: 10.1146/annurev-physiol-021115-105339. Epub 2015 Nov 19. PMID 26654352
- [Background] Laurens C, Bergouignan A, Moro C. Exercise-Released Myokines in the Control of Energy Metabolism. Front Physiol. 2020 Feb 13;11:91. doi: 10.3389/fphys.2020.00091. eCollection 2020. PMID 32116795
- [Background] Quinn A, Doody C, O'Shea D. The effect of a physical activity education programme on physical activity, fitness, quality of life and attitudes to exercise in obese females. J Sci Med Sport. 2008 Sep;11(5):469-72. doi: 10.1016/j.jsams.2007.07.011. Epub 2007 Sep 14. PMID 17869182
- [Background] Pedersen BK. The diseasome of physical inactivity--and the role of myokines in muscle--fat cross talk. J Physiol. 2009 Dec 1;587(Pt 23):5559-68. doi: 10.1113/jphysiol.2009.179515. Epub 2009 Sep 14. PMID 19752112
- [Background] Gadde KM, Martin CK, Berthoud HR, Heymsfield SB. Obesity: Pathophysiology and Management. J Am Coll Cardiol. 2018 Jan 2;71(1):69-84. doi: 10.1016/j.jacc.2017.11.011. PMID 29301630

DOCUMENTS (2):
  • Study Protocol (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT06680713/Prot_000.pdf
  • Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT06680713/ICF_001.pdf